CLINICAL TRIAL: NCT06037226
Title: A National Observation Study on Pelvic Floor Dysfunction Diseases Based on Electrophysiological Technology and a Newly Established Prevention and Treatment System in China
Brief Title: A National Observation Study on Pelvic Floor Dysfunction Diseases in China
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PekingUMCH-2021YFC20701303
Record Dates: First submitted 2023-09-08; First posted 2023-09-14 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2022-10

CONDITIONS: Pelvic Floor Dysfunction
Keywords: Pelvic floor dysfunction, postpartum women

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Postpartum pelvic floor rehabilitation — biofeedback with Pelvic floor muscle training (PFMT)

SUMMARY:
In this protocol, our team intend to conduct a nation-wide multicenter cohort research to screening for PFD symptoms in early postnatal women in China. Beside clinically significant symptoms, we will also measure the recovery trend of pelvic muscle function, aiming to determine the clinically significant alterations that are sensitive to predict the PFD risks. This is an observational prospective cohort study, following a natural regular clinical visit process. Patients will voluntarily decide whether to receive PFD related treatments and the types of treatments to adopt. Therefore, we will also be able to compare the effectiveness of treatments.

ELIGIBILITY:
Inclusion Criteria:

1. Postpartum women: 42 days+15 days after delivery
2. Age:20-45
3. Consent to participate in the research.

Exclusion Criteria:

1. Refuse gynecological and/or obstetrical examinations.
2. Diagnosed with psychiatric disorders
3. Diagnosed with other severe illnesses
4. Received pelvic floor treatments
5. Other factors that may confound with the research

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All adult women in early postnatal period, 42 days+15 days after delivery, are eligible to participate.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-02 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Urinary incontinence | 6 months
  UI will be diagnosed via gynecological examination and self-reported symptoms

SECONDARY OUTCOMES:
Pelvic organ prolapse | 6 months
  Physical examinations will be performed to diagnose the incidence and degree of organ prolapse (i.e. anterior vaginal wall prolapse, posterior vaginal wall prolapse, uterine prolapse, and vaginal apex prolapse) according to the Pelvic Organ Prolapse Quantification (POP-Q).

OTHER OUTCOMES:
Pelvic muscle function | 6 months
  In palpation, pelvic floor muscle strength will be graded based on the Oxford Muscle Scale and Electronic-muscle strength Medical Record system

IPD SHARING:
Plan to Share IPD: No